CLINICAL TRIAL: NCT05165849
Title: A Multicenter, Open-label, Phase I/Ⅱ Study to Evaluate the Safety/Tolerability, Pharmacokinetics, and Efficacy of GFS101A in Combination With Toripalimab Treating Patients With Advanced Solid Tumors
Brief Title: A Study of GFS101A in Combination With Toripalimab in Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: sponsor decided to withdraw the study
Sponsor: Zhejiang Genfleet Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFS101AX0101
Record Dates: First submitted 2021-12-06; First posted 2021-12-21 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GFS101A+Toripalimab (Experimental): Patient will be administrated with GFS101A IV in combination with Toripalimab IV. The duration of the treatment cycle is defined as 21 days.
  Interventions: Drug: GFS101A; Drug: Toripalimab

INTERVENTIONS:
Drug: GFS101A — GFS101A will be administrated intravenously Q3W.
Drug: Toripalimab — Toripalimab with fixed dose of 240 mg Q3W administered intravenously.

SUMMARY:
The purpose of this study is to evaluate the safety/tolerability, pharmacokinetics, and efficacy of GFS101A in combination with Toripalimab in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical trial, and are willing to sign informed consent forms.
2. Male or female aged from 18-75 years old (inclusive).
3. Diagnosed with histologically or cytologically confirmed advanced solid tumors.
4. Evaluable lesions defined by RECIST v1.1.
5. Eastern Cooperative Oncology Group performance status of 0 to 1.
6. Subjects or their legal representatives are able to communicate well with Investigators and are willing to comply with the protocol and complete the study.

Exclusion Criteria:

1. With clinically significant cardiac diseases
2. With clinically significant digestive disorders.
3. Other severe disease.
4. Pregnant or lactating women.
5. Other unfavorable situations for subjects to participate in the study judged by Investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Phase I：Incidence of dose limiting toxicity (DLT) events | 21days
Phase II: Overall response rate (ORR) per RECIST 1.1 | approximately 12 months after first dose